CLINICAL TRIAL: NCT03890978
Title: Improving Exclusive Breastfeeding Via Mobile Phone Text Messages: a Randomized Controlled Trial in Southern Jordan
Brief Title: Improving Exclusive Breastfeeding Via Mobile Phone Text Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Reham Mohammad Khresheh, Reham Mohammad Khresheh, Mutah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2432019
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Breastfeeding
Keywords: exclusive, breastfeeding, text messages, Jordan
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The intervention group will receive EBF promotional messages from the time of discharge until 6 months post delivery.
  Interventions: Other: promotional Exclusive breastfeeding text messages
- control (Other): the control group will receive child health care-related messages (except breastfeeding messages) from the time of discharge until 6 months post delivery.
  Interventions: Other: promotional Exclusive breastfeeding text messages

INTERVENTIONS:
Other: promotional Exclusive breastfeeding text messages — promotional Exclusive breastfeeding text messages will be send to women via mobile phone

SUMMARY:
World Health Organization (2001) recommended that infants should be exclusively breastfed for the first 6 months and could be continued in the second year of life or longer. The rate of exclusive breastfeeding (EBF) in Jordan is in progressive decline. In 2002 the EBF rate among babies less than 6 months old was 26.7% and unfortunately this rate dropped to 22% in 2007 and to 23% in 2012. In Jordan, 68% of babies receive breast milk within 24 hours of birth and the large majority continues to do so for 12.5 months, but EBF rates are very low. While health and nutrition experts recommend that introduction of complementary foods should start only when an infant is six months old, other liquids such as water, juice, and formula milk are being introduced to most Jordanian infants in the first couple of months . Thus, urgent attention is directed towards improving exclusive breastfeeding rates during the first six months of life.Despite scientific evidence concerning the benefits of breast milk, the practice of EBF is still uncommon in Jordan. Even with the consolidation of numerous strategies to promote breastfeeding and the general public health recommendation that infants should be exclusively breastfed during the first six months of life, the duration of breastfeeding in Jordan is in progressive decline and the percentage of infants exclusively breastfed for the first six months of life is still low and worrisome. A review of previous studies in Jordan, showed that most of these are descriptive studies focused on studying the factors affecting the rate of EBF and the reasons why women stop breastfeeding their children. There is no study on improving EBF for women in Jordan so far. To date there have been no interventions using mobile phones to improve breastfeeding and other feeding practices in Jordan. The aim of this research is to improve the EBF rates and duration through using a mobile phone-based EBF promotion (Text message). A randomized controlled trial with follow-up from recruitment until 6 months post-delivery will be conducted to implement EBF promotion intervention using mobile phone text messages in southern Jordan, and evaluate its impact on breastfeeding practices. The intervention group will receive EBF promotional messages and the control group will receive child health care-related messages (except breastfeeding messages) from the time of discharge until 6 months post delivery.

DETAILED DESCRIPTION:
World Health Organization (2001) recommended that infants should be exclusively breastfed for the first 6 months and could be continued in the second year of life or longer. Exclusive breastfeeding (no additional food, liquids or water) for the first six months helps protect children against diseases, supports healthy brain development and is associated with better educational achievement (World Health Organization, 2013). Breastfeeding is known to provide nutritional, immunologic, psychological, social, economic, and environmental benefits (World Health Organization, 2013, 2013b) and promote stronger attachment between mother and baby (Rapley, 2002). Evidence from the literature strongly indicate that this optimal method of infant feeding should be encouraged to ensure the best possible health outcomes for women and their children(Racine, Frick, Guthrie, & Strobino, 2009). However, few of the world's newborns, including in Jordan, are exclusively breastfed for the first six months of life.

In Jordan, religion and culture support breastfeeding, but still the breastfeeding practices are not optimal. The rate of exclusive breastfeeding (EBF) in Jordan is in progressive decline. In 2002 the EBF rate among babies less than 6 months old was 26.7% and unfortunately this rate dropped to 22% in 2007 and to 23% in 2012 (Department of Statistics 2013). In Jordan, 68% of babies receive breast milk within 24 hours of birth and the large majority continues to do so for 12.5 months, but EBF rates are very low(Department of Statistics 2013). While health and nutrition experts recommend that introduction of complementary foods should start only when an infant is six months old, other liquids such as water, juice, and formula milk are being introduced to most Jordanian infants in the first couple of months(World Health Organization, 2001). Thus, urgent attention is directed towards improving exclusive breastfeeding rates during the first six months of life.

Research studies to date examining breastfeeding practices in both developed and developing countries have found high rates of breastfeeding initiation and also that this high initiation rate is accompanied by a sharp fall in EBF in the first 6 months of life(Alzaheb, 2017; Jones, Kogan, Singh, Dee, & Grummer-Strawn, 2011). For example in Australia a high initiation rate of 92% was found for EBF from 2004 to 2005 , this rate then dropped to 71% of infants who exclusively breastfed at 1 month of age, 56% at 3 months, and 14% at 6 months (Akca, et al., 2017). Similarly, in Jordan, findings from a recent research study indicate that 51% of infants began EBF within 24 hours, falling to 47% at 1 month of age, and 33% at 6 months (Khasawneh & Khasawneh, 2017).

Significance of the study Despite scientific evidence concerning the benefits of breast milk, the practice of EBF is still uncommon in Jordan. Even with the consolidation of numerous strategies to promote breastfeeding and the general public health recommendation that infants should be exclusively breastfed during the first six months of life, the duration of breastfeeding in Jordan is in progressive decline and the percentage of infants exclusively breastfed for the first six months of life is still low and worrisome. A review of previous studies in Jordan, showed that most of these are descriptive studies focused on studying the factors affecting the rate of EBF and the reasons why women stop breastfeeding their children. There is no study on improving EBF for women in Jordan so far. To date there have been no interventions using mobile phones to improve breastfeeding and other feeding practices in Jordan. The aim of this research is to improve the EBF rates and duration through using a mobile phone-based EBF promotion (Text message).

METHODS Design A randomized controlled trial with follow-up from recruitment until 6 months post-delivery will be conducted to implement EBF promotion intervention using mobile phone text messages in southern Jordan, and evaluate its impact on breastfeeding practices. The intervention group will receive EBF promotional messages and the control group will receive child health care-related messages (except breastfeeding messages) from the time of discharge until 6 months post delivery.

Hypothesis 1- The primary hypothesis of the proposed study is: The EBF rates in the intervention group during the 6 months after delivery will increase 2- fold that of the control group.

- The secondary hypotheses are: Receiving breastfeeding promotional text messages will result in higher appropriate infant feeding practices in the intervention group compared to that of the control group.

Setting The study will be conducted at Al-Karak hospital the main governmental and teaching hospital in the southern region of Jordan. In 2016 the hospital reported that on average 2,808 births occurred, 59% were caesarean births (Ministry of Health, 2017). In this hospital, there is a higher possibility of recruiting women from a diverse range of socioeconomic backgrounds. The hospital is accredited as a baby friendly hospital initiative and follows guidelines to provide early initiation of breastfeeding. The hospital has a policy to encourage mothers to give colostrum to babies within 1 hour after birth regardless of the type of delivery.

Study population Inclusion criteria will be mothers who (1) are 18 years of age and older, (2) speak and write in Arabic language, (3) could access a mobile phone that could display Arabic language fonts,(4) express interest in breastfeeding, (5) had an uncomplicated singleton pregnancy, and who lived in an area with mobile network coverage. Exclusion criteria will be (1) Non-Arabic speaking mothers, (2) who do not express interest in breastfeeding, (3) had pregnancy complications, a multiple pregnancy, and known medical conditions including mental illness that might hinder breastfeeding.

Recruitment, Assignment, and Allocation Participant eligibility will be accessed via a hospital attendance registry (used by hospital staff) in which information such as age, address, and phone numbers are recorded. At recruitment, researcher will identify potential participants with the help of hospital nurses, explained the study, provided an information statement and consent form written in Arabic, and confirmed eligibility. If a mother agreed to participate, informed consent will be obtained, and she will be requested to complete the baseline survey questions. The participant's mobile phone will be checked for compatibility with text messages and, if needed, brief training on how to read text messages will be provided.

Eligible mothers will be randomized to the intervention or control group according to an allocation sequence that will be generated by the researcher using a computer program. Each study and group number will be kept in an opaque envelope to conceal the allocation sequence and securely stored. At recruitment, researcher sequentially will take an envelope for each consenting participant and conducted the baseline interview to collect baseline data. After the participant's information is recorded, the envelope will be opened and the group allocation will be recorded.

Blinding Because the intervention could not be blinded, bias will be minimized by ensuring both groups received messages and by not explaining in the consent and information sheets how the text messages differed between groups. The information statement that will be provided only general information that each participant could be allocated randomly into a group; will receive messages containing information on childcare, and breastfeeding practices; and that the frequency of messages could vary from 1 to 3 times per week. Research staff and interviewers (via telephone) will be blinded to each participant's group status although they might guess the group based on participants' responses. To minimize bias, we will also blind research staff to the trial aims and hypotheses.

Sample size Sample size was calculated with median effect size, 95% power, 5% alpha, and 25% expected loss at follow-up. The estimated sample size is 210 (105 per group) and the final sample size requirement will be 260 participants to allow for 25% loss at follow-up, 130 each group.

Data collection Baseline data will be collected from mothers during recruitment. Follow-up (outcome) data will be collected by monthly phone calls at 1 to 6 months post delivery.

Baseline Data Collection

1. A structured form (appendix 1) will be use to collect baseline data prior to discharge, participants will be asked to provide information on their socioeconomic status, previous pregnancies and breastfeeding history, knowledge and sources of breastfeeding information, intention to breastfeed, and intended breastfeeding patterns.
2. Also information on childbirth outcomes will be collected including type of delivery and the newborn's birth weight, sex, and perinatal outcomes.
3. Breastfeeding self efficacy will be assessed before discharge using the Arabic version breastfeeding self-efficacy scale(C. L. Dennis, 2003). The short form of the instrument, the BSES-SF, which was developed by Dennis, retains only 14 of the original 33 items and has also been shown to be a reliable (Cronbach's alpha coefficient was 0.94) and a valid measure of breast-feeding self-efficacy and to predict breast-feeding initiation, duration, and exclusivity (C. L. Dennis, 2003). The BSES-SF is made up of 14 items based on 5-point likert scale, where the mothers respond to each of the statements by checking a number from 1 to 5, whereby 1 denotes "not at all confident" and 5 denotes "very confident". All items are presented positively and begin by the idiom "I can always".

Follow-Up Data Collection Follow-up data collection will comprise feeding follow-up assessments, morbidity, breastfeeding self-efficacy Scale.

1. The feeding follow-up form (appendix 2) will be completed every month and asked if the infant is breastfed and if other liquids or foods were given in the last 24 hours and over the preceding month since the last contact (or birth for the first follow-up). Each participant will complete 6 assessments of their feeding practices, including detailed information about the different types of liquids and foods.
2. Child morbidity status (appendix 2) will be assessed when the child is 1, 3, and 5 months of age using a structured form. Child morbidity questions (ref) will be used to record whether the child has had any signs or symptoms such as fever, cough, cold, running nose, rapid breathing, and difficulty in breathing, chest in drawing, and diarrhea and dysentery. If one of these was present, duration of illness will be further explored
3. Breastfeeding self-efficacy will be collected at 1, 3, and 5 months post delivery to ascertain the mothers' confidence to breastfeed, the relationship between self-efficacy and breastfeeding duration, and whether text messages improved breastfeeding self-efficacy.

Outcome Measures The primary outcome is the rate of EBF at 1 to 6 months of the infants' age measured at monthly intervals after delivery. Secondary outcomes are median duration of EBF and rates of early initiation of breastfeeding (within 1 hour after birth); predominant breastfeeding; current breastfeeding; bottle feeding; and early introduction of solid, semisolid, or soft foods at 1 to 6 months of infant's age (measured at monthly intervals).

Data analysis Outcomes will be compared between groups using t-test for parametric data and Wilcoxon rank sum for nonparametric data.

Ethical consideration Approval to conduct the study will be obtained from the ethics committee at faculty of nursing / Mutah University and the Ministry of Health (MOH). Mothers will be informed about the study and verbal and written consent for agreement will be obtained from each mother . Mothers will be assured that participation is voluntary and they have the right to withdraw from the study at any time without giving any reason. Mothers will be assured that their information will not be recognized in any products of this research. Data will be stored on computer and accessed only by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* speak and write in Arabic language
* could access a mobile phone that could display Arabic language fonts,
* express interest in breastfeeding
* had an uncomplicated singleton pregnancy
* who lived in an area with mobile network coverage

Exclusion Criteria:

* Non-Arabic speaking mothers
* who do not express interest in breastfeeding
* had pregnancy complications, a multiple pregnancy, and known medical conditions including mental illness that might hinder breastfeeding.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 201 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
The rate of the Exclusive Breastfeeding | from birth of baby to 6 months post birth
  The primary outcome is the rate of EBF at 1 to 6 months of the infants' age measured at monthly intervals after delivery

SECONDARY OUTCOMES:
median duration of EBF | from birth of baby to 6 months post birth
  duration of exclusive breastfeeding
rates of early initiation of breastfeeding | within 1 hour after birth
  ates of early initiation of breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Khresheh, PhD, Principal Investigator — Mutah University
Locations (1):
- Ministry Of Health, Karak, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuidhail J, Al-Modallal H, Yousif R, Almresi N. Exclusive breast feeding (EBF) in Jordan: prevalence, duration, practices, and barriers. Midwifery. 2014 Mar;30(3):331-7. doi: 10.1016/j.midw.2013.01.005. Epub 2013 Feb 26. PMID 23484776
- [Background] Ahmed AH, Ouzzani M. Interactive web-based breastfeeding monitoring: feasibility, usability, and acceptability. J Hum Lact. 2012 Nov;28(4):468-75. doi: 10.1177/0890334412451869. Epub 2012 Aug 3. PMID 22864059
- [Background] Akca A, Corbacioglu Esmer A, Ozyurek ES, Aydin A, Korkmaz N, Gorgen H, Akbayir O. The influence of the systematic birth preparation program on childbirth satisfaction. Arch Gynecol Obstet. 2017 May;295(5):1127-1133. doi: 10.1007/s00404-017-4345-5. Epub 2017 Mar 16. PMID 28303340
- [Background] Al Juaid DA, Binns CW, Giglia RC. Breastfeeding in Saudi Arabia: a review. Int Breastfeed J. 2014 Jan 14;9(1):1. doi: 10.1186/1746-4358-9-1. PMID 24422991
- [Background] Alzaheb RA. Factors Influencing Exclusive Breastfeeding in Tabuk, Saudi Arabia. Clin Med Insights Pediatr. 2017 Mar 10;11:1179556517698136. doi: 10.1177/1179556517698136. eCollection 2017. PMID 28469519
- [Background] Araban M, Karimian Z, Karimian Kakolaki Z, McQueen KA, Dennis CL. Randomized Controlled Trial of a Prenatal Breastfeeding Self-Efficacy Intervention in Primiparous Women in Iran. J Obstet Gynecol Neonatal Nurs. 2018 Mar;47(2):173-183. doi: 10.1016/j.jogn.2018.01.005. Epub 2018 Feb 3. PMID 29406289
- [Background] Dennis CL, Kingston D. A systematic review of telephone support for women during pregnancy and the early postpartum period. J Obstet Gynecol Neonatal Nurs. 2008 May-Jun;37(3):301-14. doi: 10.1111/j.1552-6909.2008.00235.x. PMID 18507601
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Flax VL, Negerie M, Ibrahim AU, Leatherman S, Daza EJ, Bentley ME. Integrating group counseling, cell phone messaging, and participant-generated songs and dramas into a microcredit program increases Nigerian women's adherence to international breastfeeding recommendations. J Nutr. 2014 Jul;144(7):1120-4. doi: 10.3945/jn.113.190124. Epub 2014 May 8. PMID 24812071
- [Background] Gallegos D, Russell-Bennett R, Previte J, Parkinson J. Can a text message a week improve breastfeeding? BMC Pregnancy Childbirth. 2014 Nov 6;14:374. doi: 10.1186/s12884-014-0374-2. PMID 25369808
- [Background] Jiang H, Li M, Wen LM, Hu Q, Yang D, He G, Baur LA, Dibley MJ, Qian X. Effect of short message service on infant feeding practice: findings from a community-based study in Shanghai, China. JAMA Pediatr. 2014 May;168(5):471-8. doi: 10.1001/jamapediatrics.2014.58. PMID 24639004
- [Background] Jones JR, Kogan MD, Singh GK, Dee DL, Grummer-Strawn LM. Factors associated with exclusive breastfeeding in the United States. Pediatrics. 2011 Dec;128(6):1117-25. doi: 10.1542/peds.2011-0841. Epub 2011 Nov 28. PMID 22123898
- [Background] Jordan ET, Ray EM, Johnson P, Evans WD. Text4Baby: using text messaging to improve maternal and newborn health. Nurs Womens Health. 2011 Jun-Jul;15(3):206-12. doi: 10.1111/j.1751-486X.2011.01635.x. No abstract available. PMID 21672170
- [Background] Kannisto KA, Koivunen MH, Valimaki MA. Use of mobile phone text message reminders in health care services: a narrative literature review. J Med Internet Res. 2014 Oct 17;16(10):e222. doi: 10.2196/jmir.3442. PMID 25326646
- [Background] Khasawneh W, Khasawneh AA. Predictors and barriers to breastfeeding in north of Jordan: could we do better? Int Breastfeed J. 2017 Dec 8;12:49. doi: 10.1186/s13006-017-0140-y. eCollection 2017. PMID 29234457
- [Background] Khresheh R, Suhaimat A, Jalamdeh F, Barclay L. The effect of a postnatal education and support program on breastfeeding among primiparous women: a randomized controlled trial. Int J Nurs Stud. 2011 Sep;48(9):1058-65. doi: 10.1016/j.ijnurstu.2011.02.001. Epub 2011 Feb 24. PMID 21353220
- [Background] Odone A, Ferrari A, Spagnoli F, Visciarelli S, Shefer A, Pasquarella C, Signorelli C. Effectiveness of interventions that apply new media to improve vaccine uptake and vaccine coverage. Hum Vaccin Immunother. 2015;11(1):72-82. doi: 10.4161/hv.34313. Epub 2014 Nov 1. PMID 25483518
- [Background] Oweis A, Tayem A, Froelicher ES. Breastfeeding practices among Jordanian women. Int J Nurs Pract. 2009 Feb;15(1):32-40. doi: 10.1111/j.1440-172X.2008.01720.x. PMID 19187167
- [Background] Racine EF, Frick K, Guthrie JF, Strobino D. Individual net-benefit maximization: a model for understanding breastfeeding cessation among low-income women. Matern Child Health J. 2009 Mar;13(2):241-9. doi: 10.1007/s10995-008-0337-1. Epub 2008 Mar 21. PMID 18357417
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276